CLINICAL TRIAL: NCT02674464
Title: Comparative Effectiveness of Health System vs. Multilevel Interventions to Reduce Hypertension Disparities
Brief Title: Reducing Inequities in Care of Hypertension, Lifestyle Improvement for Everyone (RICH LIFE Project)
Acronym: RICH LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00085630; UH3HL130688 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-02-04 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Uncontrolled Hypertension
MeSH Terms: interventions — Ethnicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Plus (Active Comparator): The standard of care plus arm will include audit and feedback of blood pressure control rates at the provider level along with web-based training about: 1) barriers to blood pressure and cardiovascular disease (CVD) risk factors management in at-risk patient populations; 2) strategies to address healthcare disparities in clinical settings; and 3) appropriate blood pressure (BP) measurement techniques for all clinical staff. The Hopkins research team will help clinics develop audit and feedback mechanisms if they are lacking and will provide all blood pressure measurement and web-based training.
  Interventions: Behavioral: Provider Audit-Feedback, Stratified by Race and Ethnicity; Behavioral: Blood Pressure Measurement Standardization
- Collaborative Care/Stepped Care (CC/SC) (Experimental): The CC/SC arm includes: -BP training -Audit and feedback dashboard, data stratified by race, ethnicity, payor status -A 4 hour workshop for organizational leaders in quality improvement and disparities reduction, with follow up meetings for problem-solving and support, and web-based, patient-centered communication skills training program for providers and staff -Support and guidance in establishing collaborative care model (CCM): team-based care targeting health behaviors and medication adherence. The primary care provider (PCP), care manager, CHW, and specialists in: medication management, psychosocial/behavioral, and self-management will make up the CCM team -Community health workers (CHW) working on contextualized patient interactions focused on problem-solving skills and patient self-management. CHWs will visit their patients in their homes and communities -Provider access to on-call specialists for help with patients who do not achieve BP control under the CC/SC
  Interventions: Behavioral: Provider Audit-Feedback, Stratified by Race and Ethnicity; Behavioral: Blood Pressure Measurement Standardization; Behavioral: System Level Leadership Intervention; Behavioral: Collaborative Care Team Intervention; Behavioral: Community Health Worker Referral; Behavioral: Specialist Care Consultation

INTERVENTIONS:
Behavioral: Provider Audit-Feedback, Stratified by Race and Ethnicity — Transparent and timely access to and review of clinical performance data are among the key elements of successful improvement activities. The RICH LIFE Project provides the health systems with the logic to build practice and provider level hypertension (HTN) dashboards, support in building the dashboard, and education in utilizing the dashboard. The practice dashboard provides a display of the percentage of patients achieving BP control, defined as <140/90 mm Hg for the overall practice, while the provider dashboard provides a display of the percentage of patients achieving BP control for each provider's patient panel. Both the practice and provider Dashboards stratify hypertension performance data by race (White, non-Hispanic; Black, non-Hispanic; and All Hispanic) to help practice administration and clinicians evaluate differences between races and ethnicities in BP control rates. New reports are generated at least quarterly and will display data from the previous 3 months.
  Other Names: Stratified Hypertension Dashboard
Behavioral: Blood Pressure Measurement Standardization — All adult medicine staff at participating study practices receive standardized, evidence-based, best practices BP measurement training. Aspects of the training include proper patient preparation and positioning, how use of an automated BP measurement device, and executing a "screen and confirm" protocol when measuring patients' blood pressures.
Behavioral: System Level Leadership Intervention — This System-Level Leadership intervention aims to create a learning network through an inter-organizational approach to promote health equity and reduce CVD disparities. Elements of the system-level leadership intervention, then, include: 1) an introductory session during the kick-off event (baseline); 2) a quarterly 1 hour "content call" with a presentation on leading for equity and discussion among system-level leaders, community organization leaders, and interested practice champions in the CC/Stepped care arm conducted via conference call/webinar; and 3) monthly "coaching calls" for the system and practice level leaders, CMs, and CHWs in the CC/stepped care arm to discuss the interventions, while they are actively engaged in the intervention phase.
  Arms: Collaborative Care/Stepped Care (CC/SC)
Behavioral: Collaborative Care Team Intervention — The collaborative care intervention creates a collaborative care team that, at a minimum, consists of PCP, nurse, or social worker care manager, and community health worker. The collaborative care team develops the medical management plan in partnership with patients; 2) uses care coordination to maximize interaction of the patients' PCPs with other care providers addressing medication management, patient self-management, and psychosocial support on a regular, consistent basis; and 3) determines patient access to CHW support and subspecialty consultations.
  Other Names: Collaborative Care Model
  Arms: Collaborative Care/Stepped Care (CC/SC)
Behavioral: Community Health Worker Referral — As a "stepped up" component of the Collaborative Care Team Intervention for patients needing support in overcoming a variety of social determinants
  Arms: Collaborative Care/Stepped Care (CC/SC)
Behavioral: Specialist Care Consultation — As a "stepped up" component of the Collaborative Care Team Intervention for patients with complex medical conditions and/or patients that may not typically have access to specialist care
  Arms: Collaborative Care/Stepped Care (CC/SC)

SUMMARY:
The RICH LIFE Project is a two-armed, cluster-randomized trial, comparing the effectiveness of an enhanced standard of care arm, "Standard of Care Plus" (SCP), to a multi-level intervention, "Collaborative Care/Stepped Care" (CC/SC), in improving blood pressure control, patient activation and reducing disparities in blood pressure control among 1,890 adult patients with uncontrolled hypertension and cardiovascular disease risk factors at thirty primary care practices in Maryland and Pennsylvania. Fifteen practices randomized to the SCP arm receive standardized blood pressure measurement training, and audit and feedback of blood pressure control rates at the practice provider level. Fifteen practices in the CC/SC arm receive all the SCP interventions plus the implementation of the collaborative care model with additional stepped-care components of community health worker referrals and subspecialist curbside consults and an on-going virtual workshop for organizational leaders in quality improvement and disparities reduction. The primary clinical outcomes are the percent of patients with blood pressure <140/90 mm Hg and change from baseline in mean systolic blood pressure at 12 months. The primary patient reported outcome is change from baseline in self-reported patient activation at 12 months.

DETAILED DESCRIPTION:
The investigators refined research aim is to determine if a clinic-based collaborative care team, including a community health worker (CHW) to deliver community-based contextualized care, reduces disparities in blood pressure control rates, lowers cardiovascular disease (CVD) risk, and improves outcomes among patients with hypertension and other common comorbid conditions when compared to standard of care health system approaches to CVD risk management, including audit and feedback and staff and provider training.

Collaborative care includes care coordination and care management; regular and proactive monitoring and treatment to target specific patient needs using validated clinical tools and rating scales; and regular systematic caseload reviews by the care team and consultation with experts for patients who do not show clinical improvement. A typical collaborative care team includes the primary care provider, nurse care manager or coordinator, and other members of the clinic staff involved in patient care.

Intervention protocols are designed to address common comorbidities (diabetes, hyperlipidemia, depression and coronary heart disease), lifestyle factors (dietary intake, physical activity, and smoking) and medication adherence. The intensive intervention treats the "whole" patient, driven by individual patient goals and priorities, as opposed to the standard of care, which typically focuses on individual conditions. This proposed study responds directly to patient desires to feel more equipped to be involved in their care and manage multiple conditions that contribute to CVD. The investigators have worked successfully in the past with a broad range of stakeholders, including community members, patients, providers, and payors, and will continue to engage them through the research and dissemination process.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥21 years of age) obtaining primary care from a provider at a participating practice
2. A diagnosis of hypertension or SBP≥140mmHg or DBP≥90mmHg twice in the past year or on antihypertensive medications plus at least one of the following CVD risk factors:

   * Diabetes mellitus (fasting blood sugar> 125mg/dl or hemoglobin A1c>6.5 or on a hypoglycemic medication);
   * Dyslipidemia (LDL >130 mg/dl, HDL<40 or total cholesterol >200 or on a lipid lowering agent);
   * Coronary heart disease
   * Current tobacco smokers
   * Depression by International Classification of Disease, 9th edition (ICD-9), codes or Patient Health Questionnaire (PHQ) score >9

Exclusion Criteria:

1. Cardiovascular event (unstable angina, myocardial infarction) within the past 6 months
2. Serious medical condition which either limits life expectancy or requires active management (e.g., certain cancers)
3. Condition which interferes with outcome measurement (e.g., dialysis)
4. Pregnant or planning a pregnancy during study period. Nursing mothers would need approval from physician.
5. Alcohol or substance use disorder if not sober/abstinent for ≥30 days
6. Planning to leave clinic within 6 months or move out of geographic area within 18 months
7. Individuals with cognitive impairment or other condition which makes them unable to participate in the intervention
8. Participating in another lifestyle modification, weight reduction, or treatment trial

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1820 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Cooper, MD, MPH, Principal Investigator — Johns Hopkins University; Jill Marsteller, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarez C, Perrin N, Carson KA, Marsteller JA, Cooper LA; RICH LIFE Project Investigators. Adverse Childhood Experiences, Depression, Patient Activation, and Medication Adherence Among Patients With Uncontrolled Hypertension. Am J Hypertens. 2023 Mar 15;36(4):209-216. doi: 10.1093/ajh/hpac123. PMID 36322608
- [Derived] Alvarez C, Ibe C, Dietz K, Carrero ND, Avornu G, Turkson-Ocran RA, Bhattarai J, Crews D, Lipman PD, Cooper LA; RICH LIFE Project Investigators. Development and Implementation of a Combined Nurse Care Manager and Community Health Worker Training Curriculum to Address Hypertension Disparities. J Ambul Care Manage. 2022 Jul-Sep 01;45(3):230-241. doi: 10.1097/JAC.0000000000000422. PMID 35612394
- [Derived] Cooper LA, Marsteller JA, Carson KA, Dietz KB, Boonyasai RT, Alvarez C, Ibe CA, Crews DC, Yeh HC, Miller ER 3rd, Dennison-Himmelfarb CR, Lubomski LH, Purnell TS, Hill-Briggs F, Wang NY; RICH LIFE Project Investigators. The RICH LIFE Project: A cluster randomized pragmatic trial comparing the effectiveness of health system only vs. health system Plus a collaborative/stepped care intervention to reduce hypertension disparities. Am Heart J. 2020 Aug;226:94-113. doi: 10.1016/j.ahj.2020.05.001. Epub 2020 May 8. PMID 32526534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Using eligibility criteria, the study biostatistician screened participating health systems' electronic medical record (EMR) data to identify potentially eligible patients. Only patients seen within 6 months prior to the recruitment data pull were assessed for eligibility.
  Trained study staff recruited participants between August 1, 2017, and October 31, 2019. The baseline blood pressure measurement was included in the recruitment data.
Pre-assignment Details: Participants were considered enrolled upon completing the baseline survey. Whenever possible, trained study staff administered the baseline survey immediately after obtaining consent to participate.
Units Other Than Participants: Clusters
Groups:
- Standard of Care Plus: Practices in the Standard of Care Plus (SCP) comparator group received interventions designed to reinforce and standardize evidence-based hypertension care best practices across both intervention and comparator practices. The "plus" in the standard care arm included integration of proper BP measurement techniques, hypertension care best practices, and audit and feedback of hypertension control performance, as "usual care" at each practice. Additionally, health-system- and practice-level leaders at SCP practices participated in a system-level leadership engagement intervention consisting of quarterly, one-hour calls.
- Collaborative Care/Stepped Care (CC/SC): The intensive Collaborative Care/Stepped Care (CC/SC) arm includes all components of the SCP arm and plus the establishment of a practice-based collaborative care team with a stepped-care approach; quarterly hypertension dashboard education and training; and twice quarterly "coaching calls" for system- and practice-level leaders, care managers (CM), and community health workers (CHWs) the CC/SC arm to discuss the interventions during their active intervention phase.
  In the CC/SC approach, treatment for patients with prolonged uncontrolled hypertension is enhanced by adding a care manager and a community health worker (CHW) to deliver community-based contextualized care, or consultation with a panel of sub-specialists, or both, as necessary, to improve patient-centered outcomes and reduce disparities in hypertension control.
Period: Overall Study
Arm/Group | Standard of Care Plus | Collaborative Care/Stepped Care (CC/SC)
Started | 927; 15 Clusters (There were 15 practices in this arm. Each practice makes a cluster) | 893; 15 Clusters (There were 15 practices in the arm. Each practice makes a cluster)
6 Month Follow-up (6 month survey data collection of adverse events) | 771; 15 Clusters (10 deceased; 17 withdrew; 95 missed) | 806; 15 Clusters (2 deceased; 8 withdrew; 111 missed)
Completed (12 month follow-up (primary endpoint)) | 790; 15 Clusters | 733; 15 Clusters
Not Completed | 137; 0 Clusters | 160; 0 Clusters
Not completed — Death | 10 | 21
Not completed — Withdrawal by Subject | 24 | 44
Not completed — Lost to Follow-up | 97 | 92
Not completed — Outside survey window | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care Plus (SCP): Practices in the Standard of Care Plus (SCP) comparator group received interventions designed to reinforce and standardize evidence-based hypertension care best practices across both intervention and comparator practices. The "plus" in the standard care arm included integration of proper BP measurement techniques, hypertension care best practices, and audit and feedback of hypertension control performance, as "usual care" at each practice. Additionally, health-system- and practice-level leaders at SCP practices participated in a system-level leadership engagement intervention consisting of quarterly, one-hour calls.
- Total: Total of all reporting groups
Arm/Group | Standard of Care Plus (SCP) | Collaborative Care/Stepped Care (CC/SC) | Total
Number analyzed (Participants) | 927 | 893 | 1820
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (12.1) | 59.9 (11.7) | 60.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 534 | 547 | 1081
  Male | 393 | 346 | 739
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 130 | 42 | 172
  Not Hispanic or Latino | 797 | 851 | 1648
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 4
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 463 | 566 | 1029
  White | 359 | 279 | 638
  More than one race | 30 | 25 | 55
  Unknown or Not Reported | 74 | 19 | 93
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 927 | 893 | 1820
Education, highest degree [Count of Participants; unit: Participants]
  Less than high school diploma | 156 | 177 | 333
  High school diploma/GED | 434 | 428 | 862
  Some college | 113 | 105 | 218
  Bachelor's degree | 115 | 103 | 218
  Graduate degree | 105 | 77 | 182
  Missing (refused) | 4 | 3 | 7
Medicaid [Count of Participants; unit: Participants]
  Yes | 218 | 264 | 482
  No | 703 | 624 | 1327
  Missing | 6 | 5 | 11
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 151.9 (11.7) | 152.7 (12.9) | 152.3 (12.1)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 84.4 (11.7) | 86.6 (12.9) | 85.5 (12.3)
Diabetes [Count of Participants; unit: Participants] — Electronic medical record diagnosis
  Participants | 429 | 392 | 821
Hyperlipidemia [Count of Participants; unit: Participants] — Electronic medical record diagnosis
  Participants | 700 | 646 | 1346
Coronary heart disease [Count of Participants; unit: Participants] — Electronic medical record diagnosis
  Participants | 149 | 110 | 259
Depression [Count of Participants; unit: Participants] — Electronic medical record diagnosis
  Participants | 263 | 256 | 519
Smoker [Count of Participants; unit: Participants] | 267 | 280 | 547
Patient Activation Measure (PAM-13) [Mean (Standard Deviation); unit: score on a scale] — The Patient Activation Measure is comprised of 13 items. Insignia Health scores the 13 items on a theoretical 0-100 scale. Higher scores indicate the patient is more activated.
  score on a scale | 65.4 (16.2) | 66.7 (15.9) | 66.0 (16.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Controlled Blood Pressure
Description: Number of participants with Controlled Blood Pressure (<140/90 mm Hg).
Time Frame: 12 months
Population: We received BP data on 750 patients in the SCP arm and on 754 patients in the CC/SC arm from EMR's.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Plus (SCP) | Collaborative Care/Stepped Care (CC/SC)
Number analyzed (Participants) | 750 | 754
Participants | 462 | 442
Statistical Analysis 1: Comparison: Standard of Care Plus (SCP) vs Collaborative Care/Stepped Care (CC/SC); Test type: Superiority; p = 0.68, Generalized Estimating Equations (GEE) — The a priori threshold for statistical significance was <0.05; Assuming an exchangeable correlation structure; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.62 to 1.30] — CC/SC arm compared to the SCP arm

2. Primary Outcome: Patient Activation Measure (PAM-13)
Description: The Patient Activation Measure assesses knowledge, skills, and confidence in the management of one's health. It is comprised of 13 items and each item is on a 1-5 scale. Insignia health scores on a standardized overall score of 0-100 where higher scores indicate a better outcome.
Time Frame: Baseline, 12 months
Population: 790 patients in the SCP arm completed the follow-up survey at 12-months, but 1 patient did not complete the PAM-13 (primary patient-reported outcome) questions in the survey resulting in 789 patients in the sample. 733 patients in the CC/SC arm competed the follow-up survey at 12-months, but 2 patients did not complete the PAM-13 (primary patient-reported outcome) questions in the survey resulting in 731 patients in the sample.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard of Care Plus (SCP) | Collaborative Care/Stepped Care (CC/SC)
Number analyzed (Participants) | 789 | 731
score on a scale
  Baseline | 65.4 [63.4 to 67.4] | 66.1 [64.6 to 68.7]
  12 months | 66.7 [64.6 to 68.7] | 67.9 [65.8 to 70.0]
Statistical Analysis 1: Comparison: Standard of Care Plus (SCP) vs Collaborative Care/Stepped Care (CC/SC); Test type: Superiority; p = 0.60, Mixed Effects Regression — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-1.32 to 2.30] — CC/SC arm was compared to the SCP arm

3. Secondary Outcome: Mean Systolic Blood Pressure
Description: Mean Systolic Blood Pressure in mm Hg at baseline and 12 months.
Time Frame: Baseline, 12 months
Population: We received BP data on 750 patients in the SCP arm and on 754 patients in the CC/SC arm from EMR's.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Standard of Care Plus (SCP) | Collaborative Care/Stepped Care (CC/SC)
Number analyzed (Participants) | 750 | 754
mm Hg
  Baseline | 151.8 [150.3 to 153.3] | 152.5 [151.0 to 154.0]
  12 months | 137.1 [135.5 to 138.7] | 138.7 [137.1 to 140.2]
Statistical Analysis 1: Comparison: Standard of Care Plus (SCP) vs Collaborative Care/Stepped Care (CC/SC); Test type: Superiority; p = 0.38, Mixed Effects Regression — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-1.04 to 2.71]

4. Secondary Outcome: Mean Diastolic Blood Pressure
Description: Mean Diastolic Blood Pressure in mm Hg at baseline and 12 months.
Time Frame: Baseline, 12 months
Population: We received BP data on 750 patients in the SCP arm and on 754 patients in the CC/SC arm from EMR's.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Standard of Care Plus (SCP) | Collaborative Care/Stepped Care (CC/SC)
Number analyzed (Participants) | 750 | 754
mm Hg
  Baseline | 84.7 [82.8 to 86.5] | 86.7 [84.9 to 88.6]
  12 months | 78.9 [77.1 to 80.8] | 79.8 [77.9 to 81.7]
Statistical Analysis 1: Comparison: Standard of Care Plus (SCP) vs Collaborative Care/Stepped Care (CC/SC); Test type: Superiority; p = 0.05, Mixed Effects Regression — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.43 to 0.01] — CC/SC arm compared to SCP arm

5. Secondary Outcome: Change in Global Framingham Risk Score
Description: Clinical Outcome
Time Frame: Baseline, 12, 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Change in Mean Total Cholesterol (mg/dL)
Description: Clinical Outcome
Time Frame: Baseline, 12, 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Change in Mean LDL-C (mg/dL)
Description: Clinical Outcome
Time Frame: Baseline, 12, 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Change in Mean HDL (mg/dL)
Description: Clinical Outcome
Time Frame: Baseline, 12, 24 months
Reporting Status: Not Posted

9. Secondary Outcome: % With Controlled Total Cholesterol
Description: Clinical Outcome
Time Frame: Baseline
Reporting Status: Not Posted

10. Secondary Outcome: % With Controlled Total Cholesterol
Description: Clinical Outcome
Time Frame: 12 months
Reporting Status: Not Posted

11. Secondary Outcome: % With Controlled Total Cholesterol
Description: Clinical Outcome
Time Frame: 24 months
Reporting Status: Not Posted

12. Secondary Outcome: Change in Mean Glycosylated Hemoglobin (Hemoglobin A1c)
Description: Clinical Outcome
Time Frame: Baseline, 12, 24 months
Reporting Status: Not Posted

13. Secondary Outcome: % With Hemoglobin A1c< 7.0
Description: Clinical Outcome
Time Frame: Baseline
Reporting Status: Not Posted

14. Secondary Outcome: % With Hemoglobin A1c< 7.0
Description: Clinical Outcome
Time Frame: 12 months
Reporting Status: Not Posted

15. Secondary Outcome: % With Hemoglobin A1c< 7.0
Description: Clinical Outcome
Time Frame: 24 months
Reporting Status: Not Posted

16. Secondary Outcome: Change in Patient Assessment of Care for Chronic Conditions (PACIC-Plus)
Description: Patient Reported Outcome
Time Frame: Baseline, 12, 24 months
Reporting Status: Not Posted

17. Secondary Outcome: % With BP <140/90 mmHg
Description: Clinical Outcome
Time Frame: 24 months
Reporting Status: Not Posted

18. Secondary Outcome: % With BP <130/80 mmHg
Description: Clinical Outcome
Time Frame: 12 months
Reporting Status: Not Posted

19. Secondary Outcome: % With BP <130/80 mmHg
Description: Clinical Outcome
Time Frame: 24 months
Reporting Status: Not Posted

20. Secondary Outcome: % With BP <120/80 mmHg
Description: Clinical Outcome
Time Frame: 12 months
Reporting Status: Not Posted

21. Secondary Outcome: % With BP <120/80 mmHg
Description: Clinical Outcome
Time Frame: 24 months
Reporting Status: Not Posted

22. Secondary Outcome: Change in Medication Adherence 4-Item Scale
Description: Patient Reported Outcome
Time Frame: Baseline, 12, 24 months
Reporting Status: Not Posted

23. Secondary Outcome: Change in Depressive Symptoms Patient Health Questionnaire (PHQ) 8 Score
Description: Patient Reported Outcome
Time Frame: Baseline 12, 24 months
Reporting Status: Not Posted

24. Secondary Outcome: Change in Patient Ratings of Trust
Description: Patient Reported Outcome
Time Frame: Baseline, 12, 24 months
Reporting Status: Not Posted

25. Secondary Outcome: Change in Hypertension Knowledge and Attitudes
Description: Patient Reported Outcome
Time Frame: Baseline, 12, 24 months
Reporting Status: Not Posted

26. Secondary Outcome: Change in Health Related Quality of Life (PROMIS Global Scale)
Description: Patient Reported Outcome
Time Frame: Baseline, 12, 24 months
Reporting Status: Not Posted

27. Secondary Outcome: Change in Patient Attainment of Self-Defined Goals
Description: Patient Reported Outcome
Time Frame: Baseline, 12, 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events data were collected up to 1 year.
Arm/Group | Standard of Care Plus (SCP) | Collaborative Care/Stepped Care (CC/SC)
All-Cause Mortality (participants affected / at risk) | 21/927 | 34/893
Serious Adverse Events (participants affected / at risk) | 0/927 | 0/893
Other Adverse Events (participants affected / at risk) | 515/927 | 499/893
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Standard of Care Plus (SCP) (N=927) | Collaborative Care/Stepped Care (CC/SC) (N=893)
Self-reported stroke (Cardiac disorders) | 22/875 | 24/835
Myocardial infarction (Cardiac disorders) | 9/875 | 19/835
Fall precipitating medical treatment (General disorders) | 84/875 | 82/835
Hospitalizations (General disorders) | 227/875 | 212/835
Hypotension (Cardiac disorders) | 197/873 | 186/842 — Systolic blood pressure less than 90 mm Hg or diastolic blood pressure less than 60 mm Hg
Hypertension (Cardiac disorders) | 147/873 | 150/842 — Systolic blood pressure greater than or equal to 180 mm Hg or diastolic blood pressure greater than or equal to 110 mm Hg
Bradycardia (Cardiac disorders) | 3/873 | 0/842 — Heart rate less than 40 beats/minute
Hyponatremia (General disorders) | 6 | 12 — Serum sodium less than 130 mEq/L
Hypernatremia (General disorders) | 1 | 2 — Serum sodium greater than 150 mEq/L
Hypokalemia (General disorders) | 6 | 8 — Serum potassium less than 3.0 mEq/L
Hyperkalemia (General disorders) | 21 | 29 — Serum potassium greater than 5.5 mEq/L
Serum creatinine increase by at least 50% since previous measure (Renal and urinary disorders) | 9 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT02674464/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02674464/ICF_001.pdf